CLINICAL TRIAL: NCT01329614
Title: Effects of Nicotine Replacement and Repeated Cue Exposure on Cigarette Craving
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Columbia University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: 6001; K23DA025735 (NIH)
Record Dates: First submitted 2010-10-14; First posted 2011-04-06 (Estimated); Last update posted 2024-03-15 (Actual); Status verified 2024-03

CONDITIONS: Tobacco Use Disorder
Keywords: Tobacco; Nicotine; Cigarette
MeSH Terms: conditions — Tobacco Use Disorder | interventions — Nicotine Replacement Therapy; Nicotine; Autogenic Training

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Nicotine Replacement Therapy, 7mg dose (Experimental)
  Interventions: Behavioral: Cue Extinction Training; Drug: Nicotine Replacement Therapy; Behavioral: Cue Extinction Therapy; Behavioral: Progressive Muscle Relaxation
- Nicotine Replacement Therapy, 21mg dose (Experimental)
  Interventions: Behavioral: Cue Extinction Training; Drug: Nicotine Replacement Therapy; Behavioral: Cue Extinction Therapy; Behavioral: Progressive Muscle Relaxation
- Nicotine Replacement Therapy, Placebo (Placebo Comparator)
  Interventions: Behavioral: Cue Extinction Training; Behavioral: Cue Extinction Therapy; Behavioral: Progressive Muscle Relaxation
- Nicotine Replacement Therapy, 42mg dose (Experimental)
  Interventions: Behavioral: Cue Extinction Training; Drug: Nicotine Replacement Therapy; Behavioral: Cue Extinction Therapy; Behavioral: Progressive Muscle Relaxation

INTERVENTIONS:
Behavioral: Cue Extinction Training — Repeated exposure to cigarette cues while receiving Nicotine Replacement Therapy.
Drug: Nicotine Replacement Therapy — Study doctor applies a nicotine patch to the participant's shoulder blade. The patch dose is blinded by placement of a Bandaid over the patch itself.
  Other Names: Nicoderm CQ
  Arms: Nicotine Replacement Therapy, 21mg dose; Nicotine Replacement Therapy, 42mg dose; Nicotine Replacement Therapy, 7mg dose
Behavioral: Cue Extinction Therapy — Participant is repeatedly exposed to cigarette cues without being allowed to partake in nicotine use.
Behavioral: Progressive Muscle Relaxation — Participant relaxes muscles in her body, lead through the process using guided imagery and breathing techniques.

SUMMARY:
The purpose of this study is to determine whether Cue Extinction Training will reduce relapse rates in cigarette smokers using the patch to quit.

DETAILED DESCRIPTION:
Nicotine dependence is an important public health problem that contributes to significant morbidity and mortality in our society. Treatment efforts are hampered by high relapse rates, despite the development of somewhat effective treatment modalities, such as Nicotine Replacement Treatment (NRT). NRT, e.g. the nicotine patch, is successful in smoking cessation, compensating for nicotine withdrawal after quitting smoking.

However, relapse rates remain high even in quitters on the patch. It is thought that cravings related to smoking cues contribute to relapse in smokers on the patch who try to quit. Rational treatment approaches for nicotine dependence therefore include strategies to weaken the effect of smoking cues, e.g. cue extinction training (CET). During CET smokers are repeatedly exposed to smoking cues, in the absence of nicotine administration, and smokers report lessening of cue-induced craving (extinction). It is thought that the extinction of smoking cues will result in less control of the smoking cue over smoking behavior and lower relapse rates.

The investigators hypothesize that smoking quit rates on the patch will be higher after CET. To address our hypothesis the investigators first want to develop a proof of concept procedure that demonstrates that repeated cue exposure in the laboratory results in the lessening or 'extinction' of cue-induced craving. In addition, the investigators are interested in the contribution of nicotine withdrawal to cue-induced craving. To this end, the investigators propose to include a control group without nicotine replacement (i.e. placebo patch) that will also undergo the repeated cue exposure procedure.

This study will assess the effect of CET on subsequent craving triggered by smoking cues in cigarette-smoking volunteers. After overnight abstinence, participants will come into the lab, receive a patch (nicotine or placebo) and undergo the CET procedure and perform computer tests and fill out questionnaires.

The main goal of this project is to study the relationship between nicotine replacement, cue-extinction training and subsequent cue-induced craving. Showing the effectiveness of cue-extinction training in the proposed laboratory model will support the application of the cue-extinction procedure to improve relapse rates of nicotine replacement therapies in future clinical trials.

ELIGIBILITY:
Inclusion Criteria:

* A DSM-IV Diagnosis of nicotine dependence with physiological dependence. Smoke at least 15 cigarettes daily for two years.
* Not interested in treatment.
* Medically healthy on the basis of physical examination and medical history, vital signs, EKG and laboratory tests, with a negative pregnancy test for females.
* Able to perform study procedures.
* Males or females between the ages of 21-60 years.
* Female participants agree to use an effective method of birth control during the course of the study.

Exclusion Criteria:

* A DSM-IV diagnosis of abuse or dependence on alcohol or drugs other than nicotine.
* Current Axis I diagnosis or current treatment with psychotropic medications (within last 3 months).
* Lifetime history of schizophrenia or other psychotic disorders, bipolar disorder, or anxiety disorders.
* Seeking treatment for nicotine dependence.
* Participants on parole or probation.
* History of significant recent violent behavior.
* Unstable medical condition, Blood Pressure > 150/90, Pregnancy.
* History of allergic reaction to nicotine patch.
* Participants with significant cardiac history (i.e. angina pectoris, bypass surgery, or coronary artery disease.)

Ages: 21 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2009-10; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Galvanic Skin Response | 3 days, over the course of 4-5 weeks total.
  Measurements of Galvanic Skin Response (GSR) are taken while participant is exposed to the cue. The amount of change in GSR is used to determine CET's impact on cigarette craving.

CONTACTS AND LOCATIONS:
Overall Officials: S. Rob Vorel, MD, PhD, Principal Investigator — Columbia University
Locations (1):
- New York State Psychiatric Institute - Substance Use Research Center, New York, New York, United States